CLINICAL TRIAL: NCT03501407
Title: One-Health Approach to Identify Threat Posed by Tick-borne Pathogens Responsible of Unexplained Infectious Syndrome in Humans
Brief Title: Understanding Tick-borne Diseases
Acronym: OHTICKS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-002
Record Dates: First submitted 2018-03-30; First posted 2018-04-18 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-04

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample and skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erythema migrans: Patients for whom a diagnosis of acute phase of Lyme disease is done on the basis of the existence of an erythema migrans and a tick bite history in the days preceding the occurrence of erythema (before and after antibiotics treatment) will be recruited
  Interventions: Diagnostic Test: Blood samples; Diagnostic Test: skin biopsy
- No-erythema migrans: Patients with unspecific symptoms (the most common symptoms being:
  headache, arthralgia, myalgia, febrile episode) appearing within 3 months after a tick bite will be recruited
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — 1 or 2 blood samples will be collected from the patient.
Diagnostic Test: skin biopsy — A skin biopsy will be performed on the periphery of the erythema migrans
  Groups: Erythema migrans

SUMMARY:
Ticks are the major arthropod vectors transmitting pathogenic agents to humans and domestic animals in Europe, and currently, the incidence of tick-borne disease is rising. The most common European human tick-borne disease is Lyme borreliosis, with an estimated 90 000 new cases every year (compared to 300 000 new cases in the United States annually). This disease is initially clinically diagnosed by the presence of migrating erythema following a tick bite, which is then subsequently confirmed by serological tests. In parallel with classic Lyme borreliosis cases, tick-bitten patients can also present with polymorphic and on-specific clinical symptoms (asthenia, fever, myalgia, etc. …) for which there is no known etiological diagnosis. It is extremely difficult to determine the proportion of tick-bitten patients with these symptoms compared to patients which have actually contracted Lyme disease, although it is estimated that 50% of fevers following a tick bite have an unknown infectious origin.

Typical tick habitats are woodlands, prairies, pastures, and gardens. Ticks are extremely sensitive to environmental fluctuations, which are often brought about by human socio-economic changes, thus tick-borne diseases are excellent candidates for emergence. Consequently, it is incontestable that tickborne diseases pose a significant threat to our society. In addition to improving diagnostic techniques, one of the major hurdles relates to improving public and health professional knowledge about tick disease risk. The battle against tick-borne diseases is based on relatively simple prevention measures, and their effectiveness is immeasurably improved when citizens are more informed and involved.Therefore, a multidisciplinary project, bringing together veterinarians, doctors, scientists, and consultant sociologists has been designed to create a global "One Health" approach to tick-borne diseases. Specific scientific project objectives are to (1) detect, identify, and isolate new microorganisms-both unknown or unexpected-from patients or animals suffering from unexplainable symptoms following tick bites; (2) to demonstrate tick competence in their ability to transmit these agents; and (3) to generate concrete recommendations to improve tick-borne disease management.

ELIGIBILITY:
Inclusion Criteria for patient with an erythema migrans

* Age≥18 years
* Erythema migrans
* Registered with social security
* informed and written consent

Exclusion Criteria for patient with an erythema migrans

* Pregnant women
* Immunocompromised patients (undergoing chemotherapy, corticotherapy, or biotherapy)
* Chronic inflammatory disease
* Systemic disease

Inclusion Criteria for patient with no-erythema migrans:

* Age≥18 years
* Confirmed tick bite within the last 6 months prior to the appearance of inflammatory joint disease verified via joint imaging (MRI or ultrasound)
* and/or cerebrospinal fluid cyto-chemical anomalies (meningitis,albuminocytological dissociation)
* Registered with social security
* informed and written consent

Exclusion Criteria for patient with no-erythema migrans

* Pregnant women
* Immunocompromised patients (undergoing chemotherapy, corticotherapy, or biotherapy)
* Chronic inflammatory disease
* Systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient with and without an erythema migrans after ticks bite
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Isolate new microorganisms-both unknown or unexpected-from patients suffering from unexplainable symptoms following tick bites | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chirouze, MD, Principal Investigator — CHU BEsançon
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.citique.fr/